CLINICAL TRIAL: NCT00608517
Title: The Treatment of Hematologic Malignancies With Single or Double Umbilical Cord Blood Unit Transplantation Followed by Graft-versus-Host Prophylaxis With Tacrolimus and Mycophenolate Mofetil
Brief Title: Treatment of Single or Double Umbilical Cord Trans + Graft-versus-host Disease (GVHD) Prophylaxis w/ Tacrolimus & Mycophenolate Mofetil
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow accrual
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Brian Engelhardt, MD, Assistant Professor of Medicine; Hematologist/Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VICC BMT 0552; VU-VICC-BMT-0552; NCT00244036 (obsolete NCT alias)
Record Dates: First submitted 2008-01-31; First posted 2008-02-06 (Estimated); Results first posted 2010-11-10 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2012-05

CONDITIONS: Graft Versus Host Disease; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: graft versus host disease; accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); blastic phase chronic myelogenous leukemia; childhood acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; de novo myelodysplastic syndromes; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; myelodysplastic/myeloproliferative disease, unclassifiable; nodal marginal zone B-cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II adult non-Hodgkin lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; previously treated myelodysplastic syndromes; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; splenic marginal zone lymphoma; stage I multiple myeloma; stage II multiple myeloma; refractory multiple myeloma; stage III adult Burkitt lymphoma; stage III adult Hodgkin lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III chronic lymphocytic leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III multiple myeloma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV chronic lymphocytic leukemia; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; Philadelphia chromosome positive adult precursor acute lymphoblastic leukemia; Philadelphia chromosome positive childhood precursor acute lymphoblastic leukemia; refractory chronic lymphocytic leukemia; childhood myelodysplastic syndromes; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; adult nasal type extranodal NK/T-cell lymphoma; childhood nasal type extranodal NK/T-cell lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent adult T-cell leukemia/lymphoma
MeSH Terms: conditions — Graft vs Host Disease; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Hodgkin Disease; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Extranodal NK-T-Cell; Lymphoma, T-Cell, Cutaneous | interventions — Antilymphocyte Serum; Cyclophosphamide; fludarabine phosphate; Methylprednisolone; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pediatric Myeloablative conditioning (Experimental): Patients undergo total-body irradiation on days -7 to -4, and receive cyclophosphamide IV over 1 hour on days -3 and -2, methylprednisolone IV twice daily on days -3 to -1, and anti-thymocyte globulin IV over 4 hours on days -3 to -1.
  Interventions: Biological: anti-thymocyte globulin; Drug: cyclophosphamide; Drug: methylprednisolone; Radiation: total-body irradiation
- Adult Myeloablative conditioning (Experimental): Patients receive fludarabine phosphate IV over 30 minutes on days -6 to -4, cyclophosphamide IV over 1 hour on days -5 and -4, and undergo total-body irradiation on days -3 to -1.
  Interventions: Drug: cyclophosphamide; Drug: fludarabine phosphate; Radiation: total-body irradiation
- Reduced-intensity conditioning (Experimental): Patients receive fludarabine phosphate IV over 30 minutes on days -6 to -2 and cyclophosphamide IV over 1 hour on day -6 and undergo total-body irradiation on day -1.
  Interventions: Drug: cyclophosphamide; Drug: fludarabine phosphate; Radiation: total-body irradiation

INTERVENTIONS:
Biological: anti-thymocyte globulin — Given IV
  Other Names: ATG
  Arms: Pediatric Myeloablative conditioning
Drug: cyclophosphamide — Given IV
  Other Names: Cytoxin
Drug: fludarabine phosphate — Given IV
  Other Names: Fludara
  Arms: Adult Myeloablative conditioning; Reduced-intensity conditioning
Drug: methylprednisolone — Given IV
  Other Names: Medrol
  Arms: Pediatric Myeloablative conditioning
Radiation: total-body irradiation — Given daily for 1-4 days

SUMMARY:
RATIONALE: Giving chemotherapy and total-body irradiation before a donor umbilical cord blood transplant helps stop the growth of cancer and abnormal cells and helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving tacrolimus and mycophenolate mofetil before and after transplant may stop this from happening.

PURPOSE: To look at the ability of umbilical cord blood cells from one or two unrelated donors to serve as a source of stem cells for people needing a bone marrow transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the safety (as assessed by the day 100 non-relapse mortality) and feasibility of single or double umbilical cord stem cell transplantation in patients with hematological malignancies receiving graft-versus-host disease (GVHD) prophylaxis comprising tacrolimus and mycophenolate mofetil (MMF).

Secondary

* To assess sustained donor engraftment, neutrophil recovery, platelet recovery, incidence and severity of acute graft-versus-host disease (GVHD) and chronic GVHD, relapse rate, 100-day all-cause mortality, overall survival, and immune reconstitution after single or double umbilical cord stem cell transplantation in patients with hematologic malignancies receiving graft-versus-host disease(GVHD) prophylaxis comprising tacrolimus and mycophenolate mofetil (MMF).

OUTLINE:

* Conditioning: Patients receive myeloablative or reduced-intensity conditioning regimen according to age and prior treatment.

  * Myeloablative conditioning (pediatric patients): Patients undergo total-body irradiation on days -7 to -4, and receive cyclophosphamide IV over 1 hour on days -3 and -2, methylprednisolone IV twice daily on days -3 to -1, and anti-thymocyte globulin IV over 4 hours on days -3 to -1.
  * Myeloablative conditioning (adult patients 18-40 years old): Patients receive fludarabine phosphate IV over 30 minutes on days -6 to -4, cyclophosphamide IV over 1 hour on days -5 and -4, and undergo total-body irradiation on days -3 to -1.
  * Reduced-intensity conditioning (patients over 40 and no more than 50 years old OR deemed ineligible for above myeloablative conditioning regimen due to previous treatment): Patients receive fludarabine phosphate IV over 30 minutes on days -6 to -2 and cyclophosphamide IV over 1 hour on day -6 and undergo total-body irradiation on day -1.
* Umbilical cord blood transplantation (UCBT): All patients undergo single- or double-unit umbilical cord blood transplantation (UCBT)on day 0.
* Graft-versus-host disease prophylaxis: Patients receive tacrolimus IV continuously or orally twice daily on days -2 to 180 followed by a tapering and mycophenolate mofetil IV or orally twice daily on days 0-100 followed by a tapering over the next 3 months. Patients also receive filgrastim (G-CSF) IV or subcutaneously beginning on day 0* and continuing until blood counts recover.

NOTE: *In adult patients receiving a reduced intensity transplant, G-CSF will be started when the total white cell count falls below 2.5 x 109/L.

After completion of study treatment, patients are followed monthly for 1 year and then every 2-4 months thereafter.

ELIGIBILITY:
Patient and UCB Unit Selection:

Inclusion Criteria: General (Adults and Pediatrics)

Only one of the following should be present:

* Acute leukemia (lymphocytic or myeloid or undifferentiated or biphenotypic) in complete remission 2 or beyond
* Acute lymphocytic leukemia, Philadelphia chromosome positive in complete remission 1 or beyond
* Acute myeloid leukemia in complete remission 1 if it has evolved from a myeloproliferative disorder (MPD) or myelodysplastic syndrome (MDS).
* Acute leukemia in complete remission 1 if there is a failure to recover normal blood counts or the development of MDS following induction chemotherapy.
* Therapy related acute leukemia in complete remission 1 or beyond
* Chronic myeloid leukemia (CML) chronic phase-1 (imatinib failures, imatinib intolerance), or any CML beyond first chronic phase
* Myelodysplastic syndromes (Intermediate -1 or higher risk by IPSS)
* Therapy related MDS (irrespective of IPSS)
* Multiple myeloma must have had prior chemotherapy or autologous transplant
* Chronic lymphocytic leukemia must have failed two lines of conventional therapy but still chemosensitive to third line therapy.
* Chemosensitive Non-Hodgkin's lymphoma or Hodgkin's lymphoma in CR or PR after failing induction therapy.
* High risk acute leukemia/lymphoma eg Nk/T cell, HTLV associated leukemia/lymphoma, other T cell lymphoma/leukemia in first best response
* For patients with acute leukemia-they must be in a remission (less than 5% leukemic marrow blasts) at time of study entry.

Inclusion Criteria (Adults - 18 years or older)

* Karnofsky score of > 70%
* Estimated creatinine clearance of > 60 ml/min
* Left ventricular ejection fraction of >50%
* Pulmonary function test with DLCO, FEV1 and FVC of >60%
* Total bilirubin and SGOT of < 3.0 x upper limits of normal
* Note: Age 18- 40 years for adult myeloablative conditioning Age > 40 -50 years for adult reduced intensity conditioning

Inclusion Criteria (Pediatrics - 18 years and younger)

* Karnofsky or Lansky score of > 70%
* Estimated Creatinine clearance of > 60 ml/min
* Left ventricular ejection fraction of >50%
* Pulmonary function test with FEV1 and FVC of >60% (for patients >6 years of age)
* Total bilirubin and SGOT of < 3.0 x upper limits of normal
* Note: All pediatric patients will receive myeloablative conditioning

Inclusion Criteria - Donor Issues

* No available HLA identical or 1 antigen/allele mismatched (Class I-A, B or Class II DR locus) related donor

Inclusion Criteria: Umbilical Cord Blood Unit-HLA Typing

* At least a HLA 4/6 match (Class I-A, B by low resolution, Class II-DR by high resolution) to recipient
* For double UCB SCT each unit should be at least a 4/6 match (Class I-A,B by low resolution, Class II-DR by high resolution) to recipient, and should be at least a 4/6 match (Class I-A,B by low resolution, Class II-DR by high resolution) to each other

Inclusion Criteria: Umbilical Cord Blood Unit-Cell dose

* For Single UCB SCT: the unit will have ≥ 3.5 X 107 NC/kg of recipient body weight (For pediatric patients a cell dose ≥ 3.0 X 107 NC/kg of recipient body weight is acceptable). Recipient body weight will be determined as per standard guidelines.
* For Double UCB SCT: (done only if no single UCB unit ≥ 3.5 X 107 NC/kg of recipient body weight is available for adults, and ≥ 3.0 X 107 NC/kg of recipient body weight is available for pediatric patients )
* The larger of the two units (UCB1) will have a minimum cell dose of 2.0 X 107 NC/kg of recipient body weight. The smaller of the two units (UCB2) will have a minimum of 0.5 X 107 NC/kg of recipient body weight.

The total cell dose UCB1 + UCB2 will be ≥ 2.5 X 107 NC/kg of recipient body weight.

-Adult patients eligible for a double UCB SCT but without an appropriate second UCB unit will be enrolled in the study if their single UCB unit contains ≥ 2.5 x 107 NC/kg recipient body weight.

Exclusion Criteria

* Organ dysfunction as per standard guidelines. Unable to give informed consent (for adults only)
* Pregnant or lactating
* Sexually active individuals capable of becoming pregnant or causing a pregnancy who are unable or unwilling to use appropriate contraceptives.
* Active use of illicit drugs as evidenced by a positive toxicology screen for a substance not prescribed by a medical professional just prior to initiating the preparative regimen
* Actively smoking as evidenced by a positive nicotine screen just prior to initiating the preparative regimen
* HIV positive
* Patients with other unrelated malignancies will be excluded except:
* diagnosis of skin cancer (squamous cell or basal cell)
* diagnosis of cervical dysplasia (CIN I-III)
* any other malignancy which is currently in remission and was treated with curative intent more than 5 years preceding study entry
* In patients with secondary MDS or secondary acute leukemias-the previous non-hematopoietic neoplasm should be in remission but can be within 5 years of study entry

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2005-09; Primary Completion 2008-03 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Engelhardt, MD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (4):
- United States (4):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Veterans Affairs Medical Center - Nashville, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period = 9/23/2005 through 8/15/2008
Pre-assignment Details: A total of 7 people signed consent to take part in this study. Of those, 1 was determined to be ineligible.
Groups:
- Pediatric Myeloablative Conditioning: Patients undergo total-body irradiation on days -7 to -4, and receive cyclophosphamide intravenous (IV) over 1 hour on days -3 and -2, methylprednisolone IV twice daily on days -3 to -1, and anti-thymocyte globulin IV over 4 hours on days -3 to -1.
- Adult Myeloablative Conditioning: Patients receive fludarabine phosphate intravenous (IV) over 30 minutes on days -6 to -4, cyclophosphamide IV over 1 hour on days -5 and -4, and undergo total-body irradiation on days -3 to -1.
- Reduced-intensity Conditioning: Patients receive fludarabine phosphate intravenous (IV) over 30 minutes on days -6 to -2 and cyclophosphamide IV over 1 hour on day -6 and undergo total-body irradiation on day -1.
Period: Overall Study
Arm/Group | Pediatric Myeloablative Conditioning | Adult Myeloablative Conditioning | Reduced-intensity Conditioning
Started | 2 | 3 | 1
Completed | 1 | 3 | 1
Not Completed | 1 | 0 | 0
Not completed — Death | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pediatric Myeloablative Conditioning | Adult Myeloablative Conditioning | Reduced-intensity Conditioning | Total
Number analyzed (Participants) | 2 | 3 | 1 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 0 | 0 | 2
  Between 18 and 65 years | 0 | 3 | 1 | 4
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8 (1) | 31 (1) | 42 (1) | 31 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 3
  Male | 1 | 2 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 100-day Non-relapse Mortality
Description: Evaluate the safety (as determined by the day 100 non-relapse mortality) and feasibility of single or double umbilical cord blood (UCB)stem cell transplant (SCT) in adult or pediatric patients with hematologic malignancies receiving graft-versus-host disease (GVHD) prophylaxis with tacrolimus and mycophenolate mofetil (MMF).
Time Frame: 100 days
Measure: Number; unit: participants
Arm/Group | Pediatric Myeloablative Conditioning | Adult Myeloablative Conditioning | Reduced-intensity Conditioning
Number analyzed (Participants) | 2 | 3 | 1
participants | 1 | 0 | 0

2. Secondary Outcome: Number of Participants With Sustained Donor Engraftment of Umbilical Cord Blood Stem Cells
Description: Recovery of the neutrophil portion of white blood cells and showing complete donor cells.
Time Frame: 42 days
Population: Patients who received treatment and who did not die before day 42.
Measure: Number; unit: participants
Groups:
- Pediatric Myeloablative Conditioning: Patients undergo total-body irradiation on days -7 to -4, and receive cyclophosphamide intravenous (IV) over 1 hour on days -3 and -2, methylprednisolone IV twice daily on days -3 to -1, and anti-thymocyte globulin IV over 4 hours
Arm/Group | Pediatric Myeloablative Conditioning | Adult Myeloablative Conditioning | Reduced-intensity Conditioning
Number analyzed (Participants) | 1 | 2 | 0
participants | 1 | 1 |

3. Secondary Outcome: Number of Participants With Acute Graft-versus-host Disease (GVHD)
Description: Participants who exhibit acute GVHD.
Time Frame: 100 days
Measure: Number; unit: participants
Arm/Group | Pediatric Myeloablative Conditioning | Adult Myeloablative Conditioning | Reduced-intensity Conditioning
Number analyzed (Participants) | 2 | 3 | 1
participants | 0 | 1 | 0

4. Secondary Outcome: Number of Participants Who Relapsed at 1 Year
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Pediatric Myeloablative Conditioning | Adult Myeloablative Conditioning | Reduced-intensity Conditioning
Number analyzed (Participants) | 2 | 3 | 1
participants | 0 | 0 | 0

5. Secondary Outcome: Number of Subjects With All-cause Mortality
Description: Death from any cause at 100 days
Time Frame: at 100 days
Measure: Number; unit: participants
Arm/Group | Pediatric Myeloablative Conditioning | Adult Myeloablative Conditioning | Reduced-intensity Conditioning
Number analyzed (Participants) | 2 | 3 | 1
participants | 1 | 0 | 0

6. Secondary Outcome: Overall Survival
Description: Overall survival at 1 year
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Pediatric Myeloablative Conditioning | Adult Myeloablative Conditioning | Reduced-intensity Conditioning
Number analyzed (Participants) | 2 | 3 | 1
participants | 1 | 3 | 1

7. Secondary Outcome: Number of Participants With Chronic Graft Versus Host Disease (GVHD)
Description: As opposed to acute GVHD, which is characterized by rash, cholestasis, and enteritis, chronic GVHD is characterized by nausea, anorexia, ocular and oral sicca, and other organ involvement
Time Frame: 100 days
Measure: Number; unit: participants
Arm/Group | Pediatric Myeloablative Conditioning | Adult Myeloablative Conditioning | Reduced-intensity Conditioning
Number analyzed (Participants) | 2 | 3 | 1
participants | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Pediatric Myeloablative Conditioning | Adult Myeloablative Conditioning | Reduced-intensity Conditioning
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/3 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 2/3 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pediatric Myeloablative Conditioning (N=2) | Adult Myeloablative Conditioning (N=3) | Reduced-intensity Conditioning (N=1)
MRSE (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gram negative rods septicemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pediatric Myeloablative Conditioning (N=2) | Adult Myeloablative Conditioning (N=3) | Reduced-intensity Conditioning (N=1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Mucositis (functional/symptomatic) (Gastrointestinal disorders) | 0 (0) | 2 (4) | 0 (0)
Mucositis (clinical exam) (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Catheter-related infection Grade 3-4 neutrophils (ANC < 1.0 x 10e9/L) (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Infection with normal ANC or Grade 1-2 neutrophils (Infections and infestations) | 0 (0) | 2 (4) | 0 (0)
Infection with grade 3-4 neutrophils (ANC< 1.0 x 10e9/L) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Catheter-related infection grade 1-2 neutrophils (Infections and infestations) | 0 (0) | 1 (3) | 0 (0)
Infection with nomral ANC or grade 1-2 joint (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (5) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (9) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (5) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Cystitis (Renal and urinary disorders) | 0 (0) | 2 (4) | 0 (0)
Bladder spasms (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (3) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (2) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Abnormal PTT (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0)
Urinary bleeding (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 0 (0)
Limb pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 0 (0)
Testical pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (4) | 0 (0)
Errectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Libido (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes